CLINICAL TRIAL: NCT00215800
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled Study of the Safety and Efficacy of Poly I:Poly C12U (Ampligen®) 400 mg IV Twice Weekly Versus Placebo in Patients With Severely Debilitating Chronic Fatigue Syndrome (CFS)/Myalgic Encephalomyelitis (ME)
Brief Title: The Study of the Safety and Efficacy of Ampligen in Chronic Fatigue Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AIM ImmunoTech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMP 516
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis
Keywords: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis; CFS; Ampligen; Poly I:ploy C12U
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — poly(I).poly(c12,U)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ampligen

SUMMARY:
multi-center, double-blind, randomized, placebo-controlled study of the safety and efficacy.

DETAILED DESCRIPTION:
This study will be a prospective, double-blind, randomized, placebo-controlled, equal parallel groups study conducted at up to fifteen (15) centers to compare the safety and efficacy of Ampligen® IV versus placebo IV in 230-240 patients with CFS/ME. Patients will be randomized and stratified to receive either Ampligen® intravenously or placebo (normal saline) intravenously. Fifty percent (50%) of the patients will be treated with Ampligen® IV and 50% of the patients will be treated with placebo IV.

Patients will be studied until 64 weeks (STAGES I plus II) have passed or until: 1) removed because of toxicity, 2) they withdraw voluntarily, 3) a change in the patient's medical condition makes continued participation unsafe, 4) the patient becomes non-compliant with the requirements of the protocol or 4) the Sponsor terminates the study.

Official Title: A multi-center, double-blind, randomized, placebo-controlled study of the safety and efficacy of poly I:poly C12U (Ampligen®) 400 mg IV twice weekly versus placebo in patients with severely debilitating chronic fatigue syndrome (CFS)/myalgic encephalomyelitis (ME)

Further Study Details

Enrollment = 234: Study Completed

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of CFS, as defined by the Center for Disease Control (1988 CDC case definition) > 12 months (Appendix D).
2. Age Range: > 18 years old, < 60 years old.
3. Males or non-pregnant, non-lactating females: Females must be of non-child bearing potential (either post-menopausal for two (2) years or surgically sterile including tubal ligation) or using an effective means of contraception (birth control pills, intrauterine device, diaphragm). Females who are less than two (2) years post-menopausal, those with tubal ligations and those using contraception must have a negative serum pregnancy test within the two (2) weeks prior to the first study medication infusion. Females of child bearing potential agree to use an effective means of contraception from four (4) weeks prior to the baseline pregnancy test until four (4) weeks after the last study medication infusion.
4. A reduced quality of life as determined by a documented KPS of 40 to 60 on three (3) occasions, each at least 14 days apart, during the twelve (12) weeks immediately preceding the start of study drug infusions. The KPS must be rounded in increments of ten (10).
5. Ability to walk (minimum of 20 seconds) on the moving treadmill (grade = 0%; belt speed = 1 mph) on a minimum of two (2) occasions during the twelve (12) weeks immediately preceding study entry.
6. Laboratory documentation (baseline or historical following onset of CFS/ME) of a negative ANA or a negative anti-ds (double-stranded) DNA, a negative Rheumatoid Factor, and an erythrocyte sedimentation rate (ESR).
7. Laboratory documentation that the patient is euthyroid (patients on thyroid replacement therapy must be on a stable dose during the eight (8) week washout period) based on a thyroid profile (T4, T3, TSH, T3 uptake and Free T4 index) performed during baseline.
8. Ability to provide written informed consent indicating awareness of the investigational nature of this study.

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 234
Dates: Start 1998-12; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Strayer, MD, Study Director — AIM ImmunoTech Inc.

REFERENCES:
- [Derived] Strayer DR, Young D, Mitchell WM. Effect of disease duration in a randomized Phase III trial of rintatolimod, an immune modulator for Myalgic Encephalomyelitis/Chronic Fatigue Syndrome. PLoS One. 2020 Oct 29;15(10):e0240403. doi: 10.1371/journal.pone.0240403. eCollection 2020. PMID 33119613
- [Derived] Strayer DR, Carter WA, Stouch BC, Stevens SR, Bateman L, Cimoch PJ, Lapp CW, Peterson DL; Chronic Fatigue Syndrome AMP-516 Study Group; Mitchell WM. A double-blind, placebo-controlled, randomized, clinical trial of the TLR-3 agonist rintatolimod in severe cases of chronic fatigue syndrome. PLoS One. 2012;7(3):e31334. doi: 10.1371/journal.pone.0031334. Epub 2012 Mar 14. PMID 22431963